CLINICAL TRIAL: NCT04742543
Title: Virtual Reality During Conization of Cervix Uterus Under Local Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0097-21-TLV
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Dysplasia, Cervix
Keywords: cervical dysplasia; conization; anxiety; pain; virtual reality
MeSH Terms: conditions — Uterine Cervical Dysplasia; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: : Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality glasses (Experimental): Patients referred for conization due to cervical dysplasia under local anesthesia. In this arm , patients will be allocated to undergo the conization procedure with Virtual reality glasses on
  Interventions: Device: SootheVR: AppliedVR, Los Angeles, California a head-mounted display
- No intervention. standard treatment (No Intervention): Patients referred for conization due to cervical dysplasia under local anesthesia. In this arm , patients will be allocated to undergo the conization procedure without virtual reality glasses (no intervention)

INTERVENTIONS:
Device: SootheVR: AppliedVR, Los Angeles, California a head-mounted display — For the study group, virtual reality content will be shown to the participant for the duration of the conization procedure through a head-mounted display, RelieVRTM. The default VR content for the trial will be "swimming with dolphins" or any other content chosen by the participant
  Arms: Virtual reality glasses

SUMMARY:
To evaluate the effectiveness of virtual reality glasses as a distraction technique in the management of acute pain and anxiety during conization of cervix uterus under local anesthesia

DETAILED DESCRIPTION:
A prospective, open-label, randomized control trial in a tertiary university affiliated medical center between March 2021 to March 2023. Overall, 100 women referred for conization of cervix due to cervical dysplasia will be randomly allocated to undergo conization either with the use of virtual reality glasses (study group) or with standard treatment (control group). The primary outcome measures will include self-reported pain, anxiety scores, and vital signs as an indirect measurement of pain and anxiety, including pulse rate (PR) and respiratory rate (RR). Pain and anxiety outcomes will be measured as numeric rating scores.

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years referred for conization of cervix due to cervical dysplasia

Exclusion Criteria:

* patients under 18 years
* pregnant women

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — all patients are women referred for conization of cervix uterus due to cervical dysplasia
Enrollment: 100 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Assessments of pain through pain score parameter | 20 minutes
  Assessments of pain through pain score parameter of the NRS questionnaire. Pain will be measured using the Numeric Rating Scale (NRS) which is a 11 point scale from 0 to 10 which is a validated score of measuring pain in which 0 is no pain and 10 is the worst imaginable pain
Assessments of pain through physiological parameters | 20 minutes
  Assessments of pain through physiological parameters of pulse rate. Heart Rate will be measured using heart rate beats per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Lis Maternity Hospital, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No